CLINICAL TRIAL: NCT05564949
Title: A "Classic" Ketogenic Diet as a Complementary Therapeutic Management on Patients With High-grade Gliomas and Brain Metastases.
Brief Title: A Ketogenic Diet as a Complementary Treatment on Patients With High-grade Gliomas and Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Arezina Kasti, Registered Dietitian, MSc, PhDc, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ΕΒΔ246/14-04-2022
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Brain; Cancer
Keywords: ketogenic; diet; gliomas; metastases
MeSH Terms: conditions — Neoplasms; Glioma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Patients will adhere to a classic ketogenic diet for a period of 3 months with a possible extension depending on their compliance on the diet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Classic Ketogenic Diet (Experimental): Patients will adhere to a classic ketogenic diet for a period of 3 months with a possible extension depending on their compliance on the diet.
  Interventions: Other: CKD

INTERVENTIONS:
Other: CKD — Patients/families will meet with the study dietician to discuss the CKD, ask questions, and plan clinic visits. Training will take place about diet, meal planning, and ketones/glucose monitoring. The dietitian will follow the patient throughout treatment. Patients will measure their urine ketosis with urine test strips and capillary ketones with blood ketone meters daily, and they will complete records from the start till the end of the study. Finally, they will meet with the dietitian at follow-up visits and on an as-needed basis.

SUMMARY:
The survival interval of patients with gliomas ranges between 12 to 15 months. Recent findings revealed that dietary interventions to reduce glucose and glycolytic pathways could have a therapeutic effect. Ketosis can be an effective therapy to extend the survival of patients with gliomas.

DETAILED DESCRIPTION:
Gliomas are invasive and aggressive tumors, which derive from glial or stem cells, and after neoplastic transformation, acquire glial cell characteristics. Treatment of high-grade gliomas includes measures to relieve symptoms and eliminate or control the tumor. Surgery, radiation, and chemotherapy are the most common options. Recent findings revealed that dietary interventions to reduce glucose and glycolytic pathways could have a therapeutic effect. CKD is a restrictive therapeutic diet consisting of a 4:1 ratio of fat-to-CHO and protein. Fat provides up to 90% of the caloric intake, while overall CHO intake is less than 50 g/day. CKD reducing blood glucose levels and increasing ketone body levels stimulates biochemical changes to achieve systemic ketosis. Though, evidence for CKD in clinical practice is still limited. This study focuses on the classic ketogenic diet (CKD), adjusted for each patient's energy needs by dieticians to achieve ketosis. The primary outcome is to assess the efficacy of CKD to extend the survival of patients with high-grade gliomas and brain metastases. Historical controls will be used to compare the outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Karnofsky Performance Score of 50 or more.
* Newly diagnosed, histologically confirmed glioblastoma grade 4, or secondary metastases or progression after surgical resection, radiation and chemotherapy.
* Normal function of liver and kidneys
* Ability to sign informed consent form

Exclusion Criteria:

* Diabetes mellitus
* Life expectancy >3 months
* Inability to adhere to diet
* Inability to give informed consent form
* Cholecystectomy last 1 year (before the study entry)
* Diagnosis of genetic disorder of fat metabolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed from date of randomization until the date of death from any cause, assessed up to 36 months.

SECONDARY OUTCOMES:
Changes in brain tumor size | 2 years, Baseline, 3, 6, 12, and 24 months
  MRI (Magnetic Resonance Imaging) will be used to measure changes in tumor size (cm^2)
Time to progression | 2 years
Assessment of Quality of life using FACT-BR (version 4) survey | Baseline, 3, 6, 12 months
  50-item FACT-Br (Functional Assessment of Cancer Therapy - Brain) is a self-report and interview when applicable questionnaire used to assess quality of life, which includes domains such as Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Brain Cancer Subscale. Each of them is rated based on the Likert scale from 1 to 5.
Functional impairment will be assessed with the Karnofsky Performance Scale | Baseline, 3, 6, 12 months
  The scoring is assigned by a health professional based on the hierarchical scale: 100=normal, no evidence of disease, while 10=death. Intermediate or decimal scores can be assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Boviatsis, MD, Study Director — UNIVERSITY GENERAL HOSPITAL ATTIKON
Locations (2):
- Greece (2):
  - Arezina Kasti, Chaïdári, Athens
  - Attikon University General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas JG, Veznedaroglu E. Ketogenic Diet for Malignant Gliomas: a Review. Curr Nutr Rep. 2020 Sep;9(3):258-263. doi: 10.1007/s13668-020-00332-2. PMID 32720120
- [Background] Sargaco B, Oliveira PA, Antunes ML, Moreira AC. Effects of the Ketogenic Diet in the Treatment of Gliomas: A Systematic Review. Nutrients. 2022 Feb 27;14(5):1007. doi: 10.3390/nu14051007. PMID 35267981
- [Background] Ebrahimpour-Koujan S, Shayanfar M, Benisi-Kohansal S, Mohammad-Shirazi M, Sharifi G, Esmaillzadeh A. Adherence to low carbohydrate diet in relation to glioma: A case-control study. Clin Nutr. 2019 Dec;38(6):2690-2695. doi: 10.1016/j.clnu.2018.11.023. Epub 2018 Nov 30. PMID 30551899
- [Background] Perry A, Wesseling P. Histologic classification of gliomas. Handb Clin Neurol. 2016;134:71-95. doi: 10.1016/B978-0-12-802997-8.00005-0. PMID 26948349